CLINICAL TRIAL: NCT00436475
Title: Vitamin D and Calcium Homeostasis for Prevention of Type 2 Diabetes
Acronym: CaDDM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DK76092 (completed); R01DK076092 (NIH); DK76092
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Glucose Intolerance; Type 2 Diabetes Mellitus; Metabolic Syndrome
Keywords: Glucose intolerance; Type 2 diabetes mellitus; Metabolic syndrome
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Other): Vitamin D3 2,000 IU daily plus Calcium Carbonate 400 mg twice daily
  Interventions: Drug: Vitamin D3 2,000 IU orally once daily; Drug: Calcium Carbonate 400 mg orally twice daily
- 2 (Other): Vitamin D3 2,000 IU daily plus Calcium-Placebo twice daily
  Interventions: Drug: Vitamin D3 2,000 IU orally once daily; Drug: Calcium-Placebo
- 3 (Other): Vitamin D3-Placebo plus Calcium Carbonate 400 mg twice daily
  Interventions: Drug: Calcium Carbonate 400 mg orally twice daily; Drug: Vitamin D3-Placebo
- 4 (Other): Vitamin D3-Placebo plus Calcium-Placebo
  Interventions: Drug: Vitamin D3-Placebo; Drug: Calcium-Placebo

INTERVENTIONS:
Drug: Vitamin D3 2,000 IU orally once daily — Vitamin D3 2,000 IU orally once daily
  Arms: 1; 2
Drug: Calcium Carbonate 400 mg orally twice daily — Calcium Carbonate 400 mg orally twice daily
  Arms: 1; 3
Drug: Vitamin D3-Placebo — Vitamin D3-Placebo
  Arms: 3; 4
Drug: Calcium-Placebo — Calcium-Placebo
  Arms: 2; 4

SUMMARY:
The purpose of the randomized trial is to quantify the effect of vitamin D and calcium supplementation on beta-cell function, insulin sensitivity, glucose tolerance and systemic inflammation and other cardiometabolic outcomes in ambulatory adults at high risk for type 2 diabetes.

DETAILED DESCRIPTION:
There is animal and human observational evidence to suggest that vitamin D and calcium are important in modifying t2DM risk but there are critical gaps in our knowledge about the clinical magnitude of the association with t2DM and potential mechanisms in humans. We are conducting a randomized trial to quantify the effect of vitamin D and calcium supplementation on beta-cell function, insulin sensitivity, glucose tolerance and systemic inflammation and other cardiometabolic outcomes in ambulatory adults at high risk for t2DM. We anticipate that the research proposed in this application is significant because it will provide the basis for defining feasible nutritional interventions that promotes prevention of t2DM. Based on the results of the proposed studies and future work in this area, vitamin D and calcium supplementation can assume an important role in the treatment of t2DM and in the prevention of the disease in the 41 million Americans who are at risk of developing t2DM.

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: all ethnic groups
* Gender: men and women
* Age

  1. Lower age limit: 40 years inclusive
  2. Upper age limit: NONE
* BMI

  1. Lower BMI limit: 25 inclusive
  2. Upper BMI limit: 40 inclusive
* Glucose Intolerance / Mild Diabetes defined as

  1. Fasting glucose ≥100 mg/dl OR
  2. 2-hr glucose after OGTT ≥140 mg/dl OR
  3. 5.8 ≤ Hemoglobin A1c ≤ 7

Major Exclusion Criteria:

* Diabetes requiring pharmacotherapy
* Smoking
* Hyperparathyroidism
* Hypercalcemia (Calcium > 10.5 mg/dl)
* Kidney stone
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anastassios G Pittas, MD MS, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts-New England Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Pittas AG, Lau J, Hu FB, Dawson-Hughes B. The role of vitamin D and calcium in type 2 diabetes. A systematic review and meta-analysis. J Clin Endocrinol Metab. 2007 Jun;92(6):2017-29. doi: 10.1210/jc.2007-0298. Epub 2007 Mar 27. PMID 17389701
- [Background] Pittas AG, Harris SS, Stark PC, Dawson-Hughes B. The effects of calcium and vitamin D supplementation on blood glucose and markers of inflammation in nondiabetic adults. Diabetes Care. 2007 Apr;30(4):980-6. doi: 10.2337/dc06-1994. Epub 2007 Feb 2. PMID 17277040
- [Background] Pittas AG, Dawson-Hughes B, Li T, Van Dam RM, Willett WC, Manson JE, Hu FB. Vitamin D and calcium intake in relation to type 2 diabetes in women. Diabetes Care. 2006 Mar;29(3):650-6. doi: 10.2337/diacare.29.03.06.dc05-1961. PMID 16505521
- [Derived] Nunez Lopez YO, Pittas AG, Pratley RE, Seyhan AA. Circulating levels of miR-7, miR-152 and miR-192 respond to vitamin D supplementation in adults with prediabetes and correlate with improvements in glycemic control. J Nutr Biochem. 2017 Nov;49:117-122. doi: 10.1016/j.jnutbio.2017.08.007. Epub 2017 Aug 26. PMID 28945992
- [Derived] Alzaman NS, Dawson-Hughes B, Nelson J, D'Alessio D, Pittas AG. Vitamin D status of black and white Americans and changes in vitamin D metabolites after varied doses of vitamin D supplementation. Am J Clin Nutr. 2016 Jul;104(1):205-14. doi: 10.3945/ajcn.115.129478. Epub 2016 May 18. PMID 27194308
- [Derived] Mitri J, Dawson-Hughes B, Hu FB, Pittas AG. Effects of vitamin D and calcium supplementation on pancreatic beta cell function, insulin sensitivity, and glycemia in adults at high risk of diabetes: the Calcium and Vitamin D for Diabetes Mellitus (CaDDM) randomized controlled trial. Am J Clin Nutr. 2011 Aug;94(2):486-94. doi: 10.3945/ajcn.111.011684. Epub 2011 Jun 29. PMID 21715514

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D-Calcium: Vitamin D3 2,000 IU daily plus Calcium Carbonate 400 mg twice daily
- Vitamin D Only: Vitamin D3 2,000 IU daily plus Calcium-Placebo twice daily
- Calcium Only: Vitamin D3-Placebo plus Calcium Carbonate 400 mg twice daily
- Placebo-Placebo: Vitamin D3-Placebo plus Calcium-Placebo
Period: Overall Study
Arm/Group | Vitamin D-Calcium | Vitamin D Only | Calcium Only | Placebo-Placebo
Started | 23 | 23 | 22 | 24
Completed | 23 | 22 | 21 | 22
Not Completed | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D-Calcium | Vitamin D Only | Calcium Only | Placebo-Placebo | Total
Number analyzed (Participants) | 23 | 23 | 22 | 24 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 22 | 24 | 92
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (2) | 57 (2) | 57 (2) | 59 (2) | 57 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 10 | 13 | 47
  Male | 11 | 11 | 12 | 11 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 23 | 22 | 24 | 92

OUTCOME MEASURES:

1. Primary Outcome: Chang in Disposition Index, a Measure of Beta Cell Function
Description: Range is 0 to infinity Lower is better.
Time Frame: baseline and 4 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vitamin D-Calcium | Vitamin D Only | Calcium Only | Placebo-Placebo
Number analyzed (Participants) | 23 | 23 | 21 | 22
units on a scale | 287 (170) | 314 (183) | -122 (177) | -129 (174)

2. Secondary Outcome: Change in Hemoglobin A1c
Description: This outcome measures change in Hemoglobin A1c, a measure of glycemia
Time Frame: Baseline to 4 months
Measure: Mean (Standard Error); unit: % of hemoglobin
Arm/Group | Vitamin D-Calcium | Vitamin D Only | Calcium Only | Placebo-Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 24
% of hemoglobin | 0.05 (0.05) | 0.08 (0.05) | 0.09 (0.05) | 0.18 (0.04)

ADVERSE EVENTS:
Arm/Group | Vitamin D-Calcium | Vitamin D Only | Calcium Only | Placebo-Placebo
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/23 | 1/22 | 0/24
Other Adverse Events (participants affected / at risk) | 6/23 | 4/23 | 5/22 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D-Calcium (N=23) | Vitamin D Only (N=23) | Calcium Only (N=22) | Placebo-Placebo (N=24)
Hospitalization (General disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D-Calcium (N=23) | Vitamin D Only (N=23) | Calcium Only (N=22) | Placebo-Placebo (N=24)
Pain (General disorders) | 1 | 0 | 0 | 0
Injury (General disorders) | 1 | 1 | 0 | 0
URI (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Joint pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0
UTI (Renal and urinary disorders) | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0
Other (General disorders) | 0 | 0 | 2 | 2

LIMITATIONS AND CAVEATS:
Fewer participants than anticipated were enrolled because of reduction in budget.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No